CLINICAL TRIAL: NCT06442241
Title: A Phase I, Randomized, Observer-Blinded, Parallel-Controlled, Dose Escalation Study to Evaluate the Safety and Immunogenicity of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cell), LYB005, in Healthy Adults Aged 18 Years and Older
Brief Title: A Safety and Immunogenicity Trial of a Respiratory Syncytial Virus Vaccine, LYB005 in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYB005-CT-AUS-101
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Syncytial Virus (RSV); RSV Infection
Keywords: RSV vaccine; Virus Like Particle
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Group 1 (LYB005 low dose without adjuvant; young adults) (Experimental): Young adults (18-59 years old) will receive a single injection of low dose LYB005 (30μg) without adjuvant on Day 1.
  Interventions: Biological: LYB005 low dose without adjuvant
- Group 2 (LYB005 middle dose without adjuvant; young adults) (Experimental): Young adults (18-59 years old) will receive a single injection of middle dose LYB005 (60μg) without adjuvant on Day 1.
  Interventions: Biological: LYB005 middle dose without adjuvant
- Group 3 (LYB005 high dose without adjuvant; young adults) (Experimental): Young adults (18-59 years old) will receive a single injection of high dose LYB005 (120μg) without adjuvant on Day 1.
  Interventions: Biological: LYB005 high dose without adjuvant
- Group 4 (LYB005 low dose with adjuvant; young adults) (Experimental): Young adults (18-59 years old) will receive a single injection of low dose LYB005 (30μg) with adjuvant on Day 1.
  Interventions: Biological: LYB005 low dose with adjuvant
- Group 5 (LYB005 middle dose with adjuvant; young adults) (Experimental): Young adults (18-59 years old) will receive a single injection of middle dose LYB005 (60μg) with adjuvant on Day 1.
  Interventions: Biological: LYB005 middle dose with adjuvant
- Group 6 (LYB005 high dose with adjuvant; young adults) (Experimental): Young adults (18-59 years old) will receive a single injection of high dose LYB005 (120μg) with adjuvant on Day 1.
  Interventions: Biological: LYB005 high dose with adjuvant
- Group 7 (placebo; young adults) (Placebo Comparator): Young adults (18-59 years old) will receive a single injection of placebo on Day 1.
  Interventions: Biological: Placebo
- Group 8 (LYB005 low dose without adjuvant; older adults) (Experimental): Older adults (≥60 years old) will receive a single injection of low dose LYB005 (30μg) without adjuvant on Day 1.
  Interventions: Biological: LYB005 low dose without adjuvant
- Group 9 (LYB005 middle dose without adjuvant; older adults) (Experimental): Older adults (≥60 years old) will receive a single injection of middle dose LYB005 (60μg) without adjuvant on Day 1.
  Interventions: Biological: LYB005 middle dose without adjuvant
- Group 10 (LYB005 high dose without adjuvant; older adults) (Experimental): Older adults (≥60 years old) will receive a single injection of high dose LYB005 (120μg) without adjuvant on Day 1.
  Interventions: Biological: LYB005 high dose without adjuvant
- Group 11 (LYB005 low dose with adjuvant; older adults) (Experimental): Older adults (≥60 years old) will receive a single injection of low dose LYB005 (30μg) with adjuvant on Day 1.
  Interventions: Biological: LYB005 low dose with adjuvant
- Group 12 (LYB005 middle dose with adjuvant; older adults) (Experimental): Older adults (≥60 years old) will receive a single injection of middle dose LYB005 (60μg) with adjuvant on Day 1.
  Interventions: Biological: LYB005 middle dose with adjuvant
- Group 13 (LYB005 high dose with adjuvant; older adults) (Experimental): Older adults (≥60 years old) will receive a single injection of high dose LYB005 (120μg) with adjuvant on Day 1.
  Interventions: Biological: LYB005 high dose with adjuvant
- Group 14 (AREXVY; older adults) (Active Comparator): Older adults (≥60 years old) will receive a single injection of positive control AREXVY on Day 1.
  Interventions: Biological: Positive control

INTERVENTIONS:
Biological: LYB005 low dose without adjuvant — Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 1 (LYB005 low dose without adjuvant; young adults); Group 8 (LYB005 low dose without adjuvant; older adults)
Biological: LYB005 middle dose without adjuvant — Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 2 (LYB005 middle dose without adjuvant; young adults); Group 9 (LYB005 middle dose without adjuvant; older adults)
Biological: LYB005 high dose without adjuvant — Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 10 (LYB005 high dose without adjuvant; older adults); Group 3 (LYB005 high dose without adjuvant; young adults)
Biological: LYB005 low dose with adjuvant — Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 11 (LYB005 low dose with adjuvant; older adults); Group 4 (LYB005 low dose with adjuvant; young adults)
Biological: LYB005 middle dose with adjuvant — Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 12 (LYB005 middle dose with adjuvant; older adults); Group 5 (LYB005 middle dose with adjuvant; young adults)
Biological: LYB005 high dose with adjuvant — Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 13 (LYB005 high dose with adjuvant; older adults); Group 6 (LYB005 high dose with adjuvant; young adults)
Biological: Placebo — 0.9% sodium chloride injection. Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 7 (placebo; young adults)
Biological: Positive control — AREXVY. Dosage forms and strengths: Solution for injection. Administer a single dose (0.5 mL) as an intramuscular injection.
  Arms: Group 14 (AREXVY; older adults)

SUMMARY:
A phase 1, randomized, observer-blinded, parallel-controlled, dose escalation study in Australia will evaluate the safety and immunogenicity of the RSV vaccine candidate LYB005 with or without adjuvant in healthy adults aged 18 years and older.

DETAILED DESCRIPTION:
The study design includes an age- and dose-escalation (low/middle/high dose) in two adult age groups (young adults [18-59 years] and older adults [≥60 years]). Study will be conducted in two parts, part 1 will enrolled young adults and part 2 will enroll older adults. A sentinel dosing approach will be used for close monitoring of safety to minimize risk to participants. Participants will be divided into the sentinel cohort and the remainder of cohort. Participants in part 1 will receive of one of two RSV vaccine formulations at one of 3 antigen dose levels or placebo. Participants in part 2 will receive of one of two RSV vaccine formulations at one of 3 antigen dose levels or positive control AREXVY. Detailed characterization of safety (including safety laboratory evaluation) and immune responses will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Part 1-A male or female aged 18-59 years at screening; Part 2-A male or female aged 60 years and older at screening.
2. Written informed consent obtained from the subject before any assessment is performed.
3. Subjects who the investigator believes that they can and will comply with the requirements of the protocol. (e.g., complete the diary cards, and complete follow-up visits).
4. Subjects must have a Body Mass Index (BMI) between ≥18.0 and ≤35.0 kg/m^2 at screening.
5. Female subjects who are not pregnant or lactating. Female subjects with childbearing potential and their partners should use highly effective, medically accepted double-barrier contraception and will not have pregnancy and fertility plan and refrain from donating ovum from at least 28 days prior to study vaccination until study completion.

   * A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
   * Highly effective double-barrier contraception is defined as use of a condom AND one of the following: birth control pills (The Pill), depot or injectable birth control, intrauterine device (IUD), NuvaRing®, implantable contraception (e.g., Implanon).
   * Note: There is no contraception requirement for female subjects with non-childbearing potential (WNCBP). There is no contraception requirement for female subjects with non-childbearing potential (WNCBP) and WNCBP subjects' male partners must use a condom from study vaccination/Day 1 until study completion.
6. Males participating in this study who are involved in heterosexual sexual activity with a female partner of childbearing potential must agree to use highly effective, medically accepted double-barrier contraception (as described above) and refrain from donating sperm from at least 28 days prior to study vaccination until study completion; male participants with WNCBP partners must use a condom only from study vaccination/Day 1 until study completion.

Exclusion Criteria:

1. Tympanic temperature > 37.5°C at screening or prior to vaccination.
2. History or presence of any respiratory infection symptoms within 7 days prior to vaccination.
3. Previous vaccination against Respiratory Syncytial Virus (RSV). Planned administration of RSV vaccination during the study (including an investigational or non-registered vaccine), except for the investigational vaccine in this trial.
4. Received a live attenuated vaccine within 28 days before vaccination or received other vaccines within 14 days before vaccination.
5. Received any immunoglobulins or blood/plasma products within 3 months prior to vaccination.
6. Individuals with the following diseases: 1）Any acute disease or acute attack of chronic diseases or using antipyretic, analgesic or anti-allergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 24 h prior to enrolment; 2）Allergies to any component of the investigational vaccine; 3）Subject has any clinically significant history of allergic conditions to other vaccines; 4）History of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders (bipolar disorder, schizophrenia, etc.) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study; 5）Asplenia, or functional asplenia; 6）Congenital or acquired immunodeficiency or autoimmune disease; 7）Chronic administration (≥14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 3 months, with the exception of inhaled or topical steroids, or short-term use (<14 consecutive days) of oral corticosteroids; 8）Have severe cardiovascular diseases (cardiopulmonary disease, pulmonary edema), severe hepatic or renal diseases, and diabetes complications that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study; 9）History of severe thrombocytopenia or other coagulation disorders which may be contraindications for an IM; 10）Severe hypertension uncontrolled by medication with systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg; 11）Positive test for hepatitis C virus (HCV), hepatitis B surface antigen (HbsAg), human immunodeficiency virus (HIV) at screening.
7. Clinically significant laboratory abnormalities determined by the investigator at screening.
8. A positive urine drug test or alcohol breath test at screening or Day 1.
9. Recent participated in another clinical trial, with receipt of the investigational drug/vaccine within 30 days prior to screening. Currently participating in or those planning to participate in another clinical trial during the study.
10. Have donated blood or plasma within 2 weeks prior to screening.
11. Other conditions that may impact the subject's safety or influence the assessment of vaccine response, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Immediate AEs for 30 minutes post-vaccination | 30 mins after vaccination
  The incidence and severity of any adverse events (AEs) within 30 minutes after the vaccination
Solicited local and systemic AEs and unsolicited AEs | Within 7 days after vaccination
  The incidence and severity of any solicited local and systemic AEs and unsolicited AEs within 7 days after the vaccination
Unsolicited AEs | Within 28 days after vaccination
  The incidence and severity of any unsolicited AEs within 28 days after the vaccination
Clinically significant laboratory abnormalities | Day 4, Day 8, Day 29 and Day 91
  The occurrence of clinically significant laboratory abnormalities 3 days, 7 days, 28 days and 90 days after vaccination
Serious adverse events (SAEs) and adverse events of special interest (AESIs) | Within 6 months after the vaccination
  The incidence of any serious adverse events (SAEs) and adverse events of special interest (AESIs) within 6 months after the vaccination

SECONDARY OUTCOMES:
To observe the humoral immunity (antibodies level) of LYB005 vaccine | Day 15 and Day 29
  The geometric mean titer (GMT) of RSV A and RSV B neutralizing antibodies at 14 days and 28 days after the vaccination; the geometric mean concentration (GMC) of RSV PreF antibodies at 14 days and 28 days after the vaccination.
To observe the persistence of humoral immunity (antibodies level) of LYB005 vaccine | Day 91 and Day 181
  The GMT of RSV A and RSV B neutralizing antibodies at 3 and 6 months after the vaccination; the GMC of RSV PreF antibodies at 3 and 6 months after the vaccination
To observe the humoral immunity (increase in antibodies level) of LYB005 vaccine | Day 15 and Day 29
  The geometric mean fold rise (GMFR) of RSV A and RSV B neutralizing antibodies at 14 days and 28 days after the vaccination; the GMFR of RSV PreF antibodies at 14 days and 28 days after the vaccination.
To observe the persistence of humoral immunity (increase in antibodies level) of LYB005 vaccine | Day 91 and Day 181
  The GMFR of RSV A and RSV B neutralizing antibodies at 3 and 6 months after the vaccination; the GMFR of RSV PreF antibodies at 3 and 6 months after the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chang, M.D, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd., Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No